CLINICAL TRIAL: NCT05243108
Title: A Randomized Controlled Trial Study to Evaluated the Effect of Exogenous Nucleotides As an Anti-ageing Supplement in Older Adults (60-70 Years)
Brief Title: Targeting Aging and Promoting Longevity with Exogenous Nucleotides (TALENTs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Meihong Xu, Associate professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TALENTs
Record Dates: First submitted 2021-11-26; First posted 2022-02-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Aging
Keywords: anti-aging; DNA methylation age; Insulin Sensitivity/Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: completely randomized design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experiment designers used seed number 1234 to generate a random sequence of 120 random numbers on SAS software and divided the 120 random numbers into two groups based on the size of the random numbers. The larger number is Group A, and the smaller number is Group B. Both intervention drugs and placebos are produced by pharmaceutical companies without any labels and look exactly the same. Neither the trial designer nor the pharmacist participated in the trial. The researchers were responsible for recruiting subjects and assigning serial numbers according to inclusion criteria. Caregivers are responsible for dispensing, reviewing, and documenting medications. Investigators are responsible for measuring and filling out questionnaire items. Medical examinations and sample collection are carried out by hospital professionals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NTs Intervention group (Experimental): The subject of 1200mg has been given orally once a day for 4 months.
  Interventions: Dietary Supplement: dietary nucleotides
- placebo control group (Placebo Comparator): The ingredients, dosage, and usage are the same as experimental.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: dietary nucleotides — 1.2 g/d NTs (5 '-AMP, 5' -CMP, 5 '-GMPNa2, 5' -UMPNa2) ;
  Arms: NTs Intervention group
Dietary Supplement: placebo — placebo
  Arms: placebo control group

SUMMARY:
To investigate the effects of dietary nucleotides (NTs) as an anti-aging supplement, a clinical trial is carried as a randomized, double-blind, parallel design, placebo-controlled. A total of 120 subjects will be enrolled in the study, and they shall be randomly distributed between the two arms, NTs-treated, and placebo-control. They would be given several measurements, including physical examination, questionnaire survey, clinical and aging-related biomarkers tests at 0 (baseline), 2, and 4 months during the RCT.

DETAILED DESCRIPTION:
To explore the anti-aging effects of NTs and the regulation of aging-related diseases, this study plans to recruit 120 people as subjects and conduct randomized controlled trials with NTs as an intervention for 4 months. Based on computer-generated random numbers, participants who meet the inclusion criteria are randomly assigned equally to two groups: placebo control and nucleotide intervention groups. In this study, the specific nucleotide composition is 5'-AMP、5'-CMP、5'-GMPNa2、5'-UMPNa2 prepared according to the ratio of 16:41:19:24, which is consistent with the ratio in breast milk and meets the requirements of national infant formula addition and special medical food formula. The dose of 1.2 g/day used is currently approved as the ingredient dose of nucleotides in conventional commercially available health food products. At the 0、2 and 4 months of the study, comprehensive geriatric health assessment, aging biomarker testing and biological sample collection will be conducted. Among them, the comprehensive evaluation of elderly health status is carried out by physical examination and questionnaire survey, including physical health, physiological function, quality of life, cognitive function, psychosocial health, and other aspects of information. The physical examination involves both physical assessment and functional assessment, including body composition, neck circumference, waist circumference, hip circumference, middle arm circumference, calf circumference, BMR, grip strength, six-minute walk, intima-media thickness, subcutaneous AGEs, and spirometry. The scale includes health status, nutritional status, cognitive status, physical activity, and dietary status. Blood samples were used to detect the safety and senescence-related indicators of the subjects. The index system covers four modules and seventeen dimensions, including blood routine, blood biochemistry, inflammatory factors, immune antibodies, T lymphocyte subtypes, oxidative stress level, cancer markers, leukocyte telomere length, DNA methylation, γ-H2A. Blood samples are sequenced simultaneously for gene and transcriptome sequencing. Fecal samples are collected for metagenomic sequencing of intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

1. Male/females of 60 to 70 years of age
2. No serious physical or mental illness
3. Able to provide written Informed Consent
4. Able to follow verbal and written study directions
5. Must not be taking or be willing to take any supplements containing any form of nucleotides for one year prior to baseline and for the duration of the study.
6. Able to maintain consistent diet and lifestyle habits throughout the study
7. Willing to consume assigned supplement (NTs or placebo) for 4 months

Exclusion Criteria:

1. Participants on the current use of prescription or over-the-counter nucleotides
2. Having abnormal screening laboratory test values or other lab test result(s) that would preclude study participation in the judgment of the investigator
3. Documented presence of atherosclerotic disease and/or cardiopulmonary disease
4. History of drug or alcohol abuse
5. History of unstable depression or mental illness within the last 6 months for which the investigator believes could impact the participant's ability to comply with study requirements
6. Other diseases or medications, according to the investigator, that would interfere directly in the results of the study or jeopardize the health of the participant.
7. Currently, or within the past 30 days, enrolled in a different clinical investigation
8. Inability to provide a venous blood sample
9. Unable or unwilling to provide written informed consent for participation in the study

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
DNAmAge | Baseline、At 2 months、At 4 months
  DNA methylation clocks were assessed through whole-genome bisulfite sequencing (WGBS).The median of four principal component (PC)-corrected clocks (Horvath, Hannum, GrimAge, and PhenoAge) was chosen as the DNA methylation age outcome measure.
The length of Leukocyte telomere | Baseline、At 2 months、At 4 months
  Telomere length was quantified via quantitative PCR, using telomeric DNA amplification compared to a reference gene.

SECONDARY OUTCOMES:
glycolipid metabolic profile | Baseline、 At 2 months、 At 4 months
  fasting glucose, glycated hemoglobin, fasting insulin, HOMA-IR, triglycerides, total cholesterol, LDL-C, HDL-C
Body composition | Baseline、At 2 months、At 4 months
  BIA method - fat mass (grams), lean mass (grams) and total mass (grams).
Phenotypic Age | Baseline、 At 2 months、 At 4 months
  Phenotypic Age=141:50+ln(0.00553*ln(1-xb)). xb=-19:907-0.0336*albuminþ+0.095*creatinine+0.0195*glucose+0.0954*lnCRP-0.0120*lymphocyte percent+0.0268 mean cell volume+0.3356 red blood cell distribution width+0.00188 alkaline phosphatase+0.0554*white blood cell count+0.0804*chronological age
Spontaneous fluorescence of subcutaneous AGEs | Baseline、At 4 months
  AGEs test
Carotid thickness of intima media | Baseline、At 2 months、At 4 months
  ultrasound
The levels of MDA | Baseline、At 2 months、At 4 months
  In serum
The levels of GSH-Px | Baseline、At 2 months、At 4 months
  In serum
The levels of SOD | Baseline、At 2 months、At 4 months
  In serum
Body circumference | Baseline、At 4 months
  Measured with a soft tape - waist, hip, mid-arm, neck and calf circumference
Gait speed | Baseline、At 4 months
  6m walking time/speed test
The score of the Short Physical Performance Battery (SPPB) | Baseline、At 4 months
  The SPPB is a composite test that includes assessments of gait speed, a balance test, and a chair stand test. The maximum score is 12 points, and a score of ≤ 8 points indicates poor physical performance.
Time costs of TUG | Baseline、At 4 months
  For the Timed-Up and Go test, individuals are asked to rise from a standard chair, walk to a marker 3 m away, turn around, walk back and sit down again.
Grip strength | Baseline、At 4 months
  Calibrated handheld dynamometer.
Pittsburgh sleep quality index (PSQI) | Baseline、 At 4 months
  Items are categorized into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The possible score range for each component is 0 (no difficulty) to 3 (severe difficulty). The seven component scores are summed to produce a global score; higher scores represent poorer subjective sleep quality.
Score of Montreal Cognitive Assessment (MoCA) | Baseline、At 4 months
  Scores range from 0-30 (+1 for 12 or fewer years of education); a score of 26 or higher indicates normal cognitive functioning, while a score of 25 or lower indicates impaired functioning.
The levels of TNF-α in serum | Baseline、 At 2 months、 At 4 months
  Suspension array
The levels of IL-1 in serum | Baseline、 At 2 months、 At 4 months
  Suspension array
The levels of IL-6 in serum | Baseline、 At 2 months、 At 4 months
  Suspension array
The levels of ICAM-1 in serum | Baseline、 At 2 months、 At 4 months
  Suspension array
Methylation damage | Baseline、 At 4 months
  Blood sample
The level of telomere repeat binding factors-1 (TRF-1) | Baseline、 At 4 months
  Blood sample
T lymphocyte subsets | Baseline、 At 2 months、 At 4 months
  CD3+, CD4+, CD8+ were analyzed using flow cytometry
γH2AX | Baseline、 At 2 months、 At 4 months
  Phosphorylated histone H2AX (p-H2AX) was measured via ELISA

OTHER OUTCOMES:
Gut microbiota | Baseline、At 4 months
  Total bacterial DNA was extracted from fecal samples, followed by 16S-targeted amplification, high-throughput sequencing, species annotation and abundance analysis to describe the intestinal microecological structure and diversity of the subjects
Scores of Quality of life | Baseline、At 4 months
  Quality of life was measured 36-Item Short Form Survey (SF-12) questionnaire. The items are grouped into eight domain scores: physical functioning, role limitations due to physical health, pain, general health, energy, social functioning, role limitations due to emotional problems and emotional well-being. Domain scores can be collapsed to a physical component summary Physical health (PCS) and a mental component summary Mental health (MHS). Each score ranges from 0 to 100, with higher values representing the better self-perceived health-related quality of life.
Dietary intake | Baseline、 At 4 months
  Dietary intake was assessed using a combination of the 24-hour dietary record (24HR) method and the Food Frequency Questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Meihong Xu, Assis prof., Principal Investigator — Peking University
Locations (1):
- Talents project team, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang S, Song L, Fan R, Chen Q, Fu R, You M, Wu Y, Cai M, Li Y, Xu M. Nucleotides as an Anti-Aging Supplementation in Older Adults: A Randomized Controlled Trial (TALENTs study). Adv Sci (Weinh). 2025 Sep;12(33):e2417728. doi: 10.1002/advs.202417728. Epub 2025 May 28. PMID 40433895